CLINICAL TRIAL: NCT03543969
Title: Pilot Study of Adaptive BRAF-MEK Inhibitor Therapy for Advanced BRAF Mutant Melanoma
Brief Title: Adaptive BRAF-MEK Inhibitor Therapy for Advanced BRAF Mutant Melanoma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19441
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Melanoma (Skin); Skin Cancer; Skin Melanoma; Skin Carcinoma
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — encorafenib; binimetinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: BRAF-MEK Inhibitor Therapy (Experimental): Participants will receive 450 mg Encorafenib daily, along with 45 mg Binimetinib twice daily and 240 mg Nivolumab IV every 2 weeks.
  Interventions: Drug: Encorafenib; Drug: Binimetinib; Drug: Nivolumab
- Arm B (Active Comparator): Participants will receive 240 mg Nivolumab IV every 2 weeks
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Encorafenib — 450 mg encorafenib daily by mouth
  Other Names: BRAFTOVI; BRAF/MEK-inhibitor
  Arms: Arm A: BRAF-MEK Inhibitor Therapy
Drug: Binimetinib — 45 mg binimetinib daily by mouth
  Other Names: MEKTOVI; BRAF/MEK-inhibitor
  Arms: Arm A: BRAF-MEK Inhibitor Therapy
Drug: Nivolumab — 240 mg Nivolumab IV every 2 weeks
  Other Names: Opdivo

SUMMARY:
This pilot early phase I trial studies how well encorafenib, binimetinib, and nivolumab work in treating patients with BRAF mutant stage IIIC-IV melanoma. Encorafenib and binimetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with nivolumab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Giving encorafenib, binimetinib, and nivolumab may kill more tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or above
* Subjects must have cytologically or histologically-confirmed unresectable melanoma that harbors a BRAF V600E mutation determined by pyrosequencing assay or equivalent genotyping assay in a Clinical Laboratory Improvement Act (CLIA) certified laboratory, meeting one of the following American Joint Committee on Cancer (AJCC) (8th edition) staging criteria:
* AJCC stage IV
* AJCC stage IIIC or IIID with unresectable nodal/locoregional involvement
* Subjects must have baseline plasma ctDNA >= 0.5 copy/ul at time of study enrollment
* Hemoglobin >= 8.0 g/dL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 75,000/mcL
* Total bilirubin =< 2 institutional upper limit of normal (ULN), unless suspected Gilbert's syndrome
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional ULN (in participants with liver metastases =< 5 x ULN)
* Creatinine =< 2.0 institutional ULN
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Negative serum pregnancy test within 7 days prior to commencement of dosing in premenopausal women. Women of non-childbearing potential may be included without serum pregnancy test if they are either surgically sterile or have been postmenopausal for >= 1 year
* Fertile men and women must use an effective method of contraception during treatment and for at least 6 months after completion of treatment as directed by their physician. (NOTE: Patients must agree to not use hormonal contraceptives, as encorafenib can result in decreased concentration and loss of efficacy.)
* Patients on non-biologic disease modifying agents (e.g. methotrexate) or patients on corticosteroids =< 10 mg prednisone daily or equivalent are permitted to enroll
* Patients must not have had grade 3 or 4 immune-related adverse events on nivolumab that required more than 12 weeks of immune suppression with corticosteroids
* No anti-PD-1/PD-L1 or BRAF/MEK inhibitor therapy in the metastatic setting is allowed; these treatments are allowed if given in neoaduvant or adjuvant setting > 24 weeks ago. Prior radiation therapy is permitted. All adverse events associated with prior systemic therapy or radiation therapy must have resolved to =< grade 1 prior to start of study
* Subjects must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1

Exclusion Criteria:

* Female subjects who are pregnant, intend to become pregnant or are nursing
* Patients previously treated with BRAF/MEK inhibitor or anti-PD-1/PD-L1 therapy in the metastatic setting
* Uncontrolled intercurrent illness including, but not limited to, serious infection. Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants must be class 2B or better
* Patients with known human immunodeficiency virus (HIV)-infection are eligible providing they are on effective anti-retroviral therapy and have undetectable viral load at their most recent viral load test and within 90 days prior to randomization
* Patients with untreated or uncontrolled brain metastases. Patients with asymptomatic brain metastases which have been previously treated (with locoregional treatment such as radiation or surgery) and are clinically stable (i.e. not requiring corticosteroids) at the time of study start will be eligible
* Previous malignancy is not an exclusion provided that the other malignancy is considered under control, patient is not on concomitant anti-cancer drug therapy, and target lesions from melanoma are clearly defined for response assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
8 Week Completion Rate | At the end of the first 8 week treatment period
  Number of participants who reach 8 weeks with the prescribed on/off schedule without progression of disease. Progression as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

SECONDARY OUTCOMES:
Time to Treatment Failure | Up to 5 years
  Time to treatment failure, defined as the time from the day of first dose of study drugs to the first day of treatment with another regimen or with the same regimen in a non-adaptive fashion.
Objective Tumor Response Rate | Up to 5 years
  Number of participants with tumor response. Response according to RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Eroglu, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States